CLINICAL TRIAL: NCT04280497
Title: A Multicentre Concealed-Allocation Multi-arms Blinded Randomized Controlled Trial to Identify the Best Sepsis Population for Corticotherapy
Brief Title: Rapid Recognition of Corticosteroid Resistant or Sensitive Sepsis
Acronym: RECORDS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Versailles Saint-Quentin-en-Yvelines University (Other); Université Paris-Saclay (Other); Paris 12 Val de Marne University (Other); Commissariat A L'energie Atomique (Other Government); Beckman Coulter, Inc. (Industry); Lumedix (Unknown); Elice (Unknown); Biothelis (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APHP191110; 2020-000296-21 (EudraCT Number)
Record Dates: First submitted 2020-02-17; First posted 2020-02-21 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Sepsis
Keywords: Sepsis; Corticosteroid; intensive care unit; CS-resistant Sepsis; CS-sensitive Sepsis
MeSH Terms: conditions — Sepsis | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (12):
- Biomarker CIRCI neg: Corticosteroid arm (Experimental): Hydrocortisone plus fludrocortisone as treatment: hydrocortisone hemisuccinate and 9 alpha fludrocortisone as experimental treatment.
  Interventions: Drug: Administration procedures
- Biomarker CIRCI neg: Placebo arm (Placebo Comparator): Placebo: hydrocortisone placebo and 9 alpha fludrocortisone placebo as placebo treatment.
  Interventions: Drug: Administration procedures
- Biomarker endocan: Corticosteroid arm (Experimental): Hydrocortisone plus fludrocortisone as treatment: hydrocortisone hemisuccinate and 9 alpha fludrocortisone as experimental treatment.
  Interventions: Drug: Administration procedures
- Biomarker endocan: Placebo arm (Placebo Comparator): Placebo: hydrocortisone placebo and 9 alpha fludrocortisone placebo as placebo treatment.
  Interventions: Drug: Administration procedures
- Biomarker GILZ: Corticosteroid arm (Experimental): Hydrocortisone plus fludrocortisone as treatment: hydrocortisone hemisuccinate and 9 alpha fludrocortisone as experimental treatment.
  Interventions: Drug: Administration procedures
- Biomarker GILZ: Placebo arm (Placebo Comparator): Placebo: hydrocortisone placebo and 9 alpha fludrocortisone placebo as placebo treatment.
  Interventions: Drug: Administration procedures
- Biomarker CPD: Corticosteroid arm (Experimental): Hydrocortisone plus fludrocortisone as treatment: hydrocortisone hemisuccinate and 9 alpha fludrocortisone as experimental treatment.
  Interventions: Drug: Administration procedures
- Biomarker CPD: Placebo arm (Placebo Comparator): Placebo: hydrocortisone placebo and 9 alpha fludrocortisone placebo as placebo treatment.
  Interventions: Drug: Administration procedures
- Biomarker Transcriptomic SRS: Corticosteroid arm (Experimental): Hydrocortisone plus fludrocortisone as treatment: hydrocortisone hemisuccinate and 9 alpha fludrocortisone as experimental treatment.
  Interventions: Drug: Administration procedures
- Biomarker Transcriptomic SRS: Placebo arm (Placebo Comparator): Placebo: hydrocortisone placebo and 9 alpha fludrocortisone placebo as placebo treatment.
  Interventions: Drug: Administration procedures
- Biomarker Endotype B: Corticosteroid arm (Experimental): Hydrocortisone plus fludrocortisone as treatment: hydrocortisone hemisuccinate and 9 alpha fludrocortisone as experimental treatment.
  Interventions: Drug: Administration procedures
- Biomarker Endotype B: Placebo arm (Placebo Comparator): Placebo: hydrocortisone placebo and 9 alpha fludrocortisone placebo as placebo treatment.
  Interventions: Drug: Administration procedures

INTERVENTIONS:
Drug: Administration procedures — Hydrocortisone hemisuccinate / hydrocortisone placebo will be given as 50 mg intravenous bolus every 6 hours;
  9 alpha fludrocortisone / 9 alpha fludrocortisone placebo will be given as a 50 μg tablet via a nasogastric tube once per day in the morning.
  Study drugs will be started immediately after randomization (day 0 of the study), until discharge from ICU for a maximal duration of 7 days. Study drugs will be stopped without tapering off.

SUMMARY:
Main objective and primary endpoint: To compare the effect hydrocortisone plus fludrocortisone vs. placebo on a composite of death or persistent organ dysfunction - defined as continued dependency on mechanical ventilation, new renal replacement therapy, or vasopressors - assessed at 90 days on intensive care unit (ICU) adults and having different biological profiles for immune responses and corticosteroids bioactivity.

Secondary objectives and endpoints:

* Mortality and health-related quality of life at 6 months;
* Daily organ function (SOFA score days 1, 2, 3, 4, 7, 10, 14, 28, and 90);
* Daily secondary infections (up to 90 days)
* Daily blood and urinary levels of glucose, sodium and potassium (up to 28 day)
* Daily gastroduodenal bleeding (up to 28 day)
* Daily cognitive function and muscles' strength (days 1 to 28, 90 and 180 days).

DETAILED DESCRIPTION:
The potential benefits of a lower dose ( ≤ 400 mg of hydrocortisone or equivalent per day), and a longer duration at full dose ( ≥ three days) of treatment, have been investigated in numerous randomized controlled trials over the past three decades. In the past two years, guidelines for clinical practices about corticosteroids use in sepsis have been released. All but one of the guidelines, recommended against the use of corticosteroids in sepsis, except in patients with septic shock and poorly responsive to fluid replacement and vasopressor therapy. Some guidelines suggested that corticosteroids should be given as a continuous infusion rather than intermittent boluses.

Corticosteroids survival benefit is not affected by age, gender, disease severity, type of infection, source of infection, or type of pathogens. There is currently no diagnostic test for CS sensitivity/resistance in sepsis. The scientific community is competing to identify markers delineating between patients who draw survival benefit from corticosteroids (CS-sensitive sepsis) and those who may be harmed (CS-resistant sepsis). In sepsis, the deregulated response may result in systemic inflammation and organs damage, or immune paresis and secondary infections. Obviously, patients with systemic inflammation may benefit from CS whereas those with immune paresis may deteriorate. The study team had have looked for an interaction between survival in response to corticosteroids and the presence of CIRCI according to the ACTH test results (cortisol increment of less than 9µg/dL). The benefits from corticosteroids were more important in patients with CIRCI in the Ger-Inf-05 trial but not in the APROCCHS trial. Thus, current sepsis guidelines suggest that the ACTH test may not reliably guide the use of corticosteroids. Indeed, this test provides information neither on corticosteroids bioactivity nor on patient's immune status, when this information should precede any corticotherapy. Recent studies suggested that a transcriptomic signature based on 100 genes may identify a subset of paediatric sepsis that had increased risk of death when exposed to corticosteroids. Another study found transcriptomic based sepsis response signatures (SRS) associated with immune paresis (SRS1) or with systemic inflammation (SRS 2). In this study, patients with a SRS 2 transcriptomic signature had significantly higher mortality when treated with hydrocortisone. Thus, we have started exploring the mechanisms of sensitivity/resistance to corticosteroids in sepsis, namely by investigating endocan, as a surrogate of patient's inflammatory status, and GILZ expression as a marker of corticosteroids bioactivity.

This is a new multicentre concealed-allocation multi-arms, parallel-group, adaptive blinded randomized controlled trial. The overall objective of the trial is to determine whether different signatures of immune status and/or corticosteroids biological activity influence the responses to hydrocortisone plus fludrocortisone of adults with sepsis. To remain pragmatic, this trial has broad eligibility criteria and includes all patients admitted to the ICU with a primary diagnosis of sepsis. Patients will be randomly assigned to hydrocortisone plus fludrocortisone or placebo for 7 days, targeting 1800 patients with full follow-up up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patient ≥18 years old;
2. Admitted to ICU with proven or suspected infection as the main diagnosis;
3. Community acquired pneumonia related sepsis or vasopressors dependency (norepinephrine, epinephrine, vasopressin, dopamine, phenylephrine) or septic shock (vasopressor to maintain mean blood pressure of at least 65 mmHg and lactate levels above 2 mmol/l) or acute respiratory distress syndrome (ARDS: a- acute onset, i.e. within one week of an apparent clinical insult and with progression of respiratory syndrome, b- bilateral opacities on chest imaging not explained by other pulmonary pathologies, e.g. pleural effusion, atelectasis, nodules etc, c- no evidence for heart failure or volume overload, d- PaO2/FiO2 ≤ 300 mm Hg, - PEEP ≥ 5 cm H2O;
4. Patients who have been tested for one or more RECORDS specific biomarkers:

   1. CIRCI
   2. Endocan
   3. GILZ
   4. DUSP-1
   5. MDW
   6. lymphopenia
   7. Transcriptomic SRS2
   8. Endotype B
   9. PCR COVID-19
   10. PCR Influenza
   11. PCR other respiratory virus
   12. Cutaneous vasoconstrictor response to glucocorticoids
5. Patient who has signed an informed and written consent whevener he/she is able of consent, if not, if not ascent from his/her representant whenever he/she is present at time of screening for inclusion;
6. Patient affiliated to a social security system or to an universal health coverage (Couverture Maladie Universelle (CMU) in France;
7. Patient under guardianship or curatorship will be included;
8. Patient in case of simple emergency (legal definition) will be included;
9. Patients managed with covid 19 and having biological samples available.

Exclusion Criteria:

1. Pregnancy;
2. Expected death or withdrawal of life-sustaining treatments within 48 hours;
3. Previously enrolled in this study
4. Formal indication for corticosteroids according to most recent international guidelines
5. Vaccination with live virus within past 6 months
6. Hypersensitivity to hydrocortisone or fludrocortisone or (microsined betamethasone dipropionate*) or any of their excipients (spc)
7. Women of childbearing potential not using contraception
8. Nursing women * For patients included in this stratum, if applicable, do not apply the cream to an infected or ulcerated area

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1800 (Estimated)
Dates: Start 2020-04-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
3-month mortality | Daily up to 3 months
  Patient's vital status.
Persistent organ dysfunction | At baseline, 1 month and 3 months
  Persistent organ dysfunction (defined as continued dependency on mechanical ventilation, renal replacement therapy, or vasopressors) and with SOFA score ≤6 up to 90 days.

SECONDARY OUTCOMES:
Mortality at 7, 14, 28 day and 6 months | at 7, 14, 28 day and 6 months
  Patient's vital status.
Vasopressor free days | through study completion, an average of 6 month
  defined as the number of days with permanent hemodynamic stability in the absence of any vasopressor agent, norepinephrine, phenylephrine, epinephrine, dopamine, vasopressine or its analogs, and soever. When a patient will die on vasopressor therapy, the corresponding vasopressor free day will be 0.
Mechanical ventilation free days | through study completion, an average of 6 month
  defined as the number of days with permanent appropriate oxygenation while the patients is extubated and breathing spontaneously, i.e. no need for non invasive ventilation, high flow oxygen or CPAP. Other uses of non-invasive ventilation (e.g., chronic night-time use for chronic obstructive pulmonary disease) are not counted. When a patient will die on mechanical ventilation or will be discharge home on mechanical ventilation, the corresponding mechanical ventilation free day will be 0.
Organ dysfunction free days | through study completion, an average of 6 month
  Organ function (including renal function) will be assessed by the SOFA score (Vincent 1996). Organ dysfunction will be defined by a SOFA score of > 6 (Annane 2018). Organ dysfunction free days are defined by the number of days with os total SOFA score of 6 or less. When a patient will die on vasopressor therapy, the corresponding vasopressor free day will be 0.
HRQoL in 6-month survivors assessed by the EuroQol-5D (EQ-5D) | at 1, 28, 90 day and 6 months
  This questionnaire is a standardised measure of health status developed to provide a simple, generic measure of health for clinical and economic appraisal. It is made up for two components; health state description and evaluation. The health status is measured in terms of five dimensions; mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. In evaluation part, the respondents evaluate their overall health status using the visual analogue scale.
Proportion of patients with a decision to withhold and/or withdraw active treatments | through study completion, an average of 6 month
ICU and hospital length of stay | through study completion, an average of 6 month
Rate of re-admission to the ICU during the 180 days after randomization | through study completion, an average of 6 month
Safety endpoints: proportion of patients affected by any serious adverse events | up to 90 days
  Serious adverse events associated with corticosteroids, among the following: hospital-acquired infections, hyperglycemia, hypernatremia, neurological disorders (coma, stroke or muscle weakness, as defined below) during the 90 days after randomization.
Coma | up to 90 days
  Coma will be defined as a Glasgow coma score < 8
Neurologic sequelae | up to 90 days
  Neurologic sequelae will be assessed according to the score on the Muscular Disability Rating Scale (MDRS), with a score of 1 indicating no deficit, 2 minor deficit with no functional disability, 3 distal motor deficit, 4 mild-to-moderate proximal motor deficit, and 5 severe proximal motor deficit.
Proportion of patients affected by hospital-acquired infections | up to 90 days
  Proportion of patients affected by hospital-acquired infections (CTINILS. Définition des infections associées aux soins. 2007, (document in french)).
Number of episodes of hyperglycemia | daily during ICU stay or up to 90 days
  Number of episodes of hyperglycemia (blood glucose levels >150mg/dl) during ICU stay (or up to day 90, whichever occurs first)
Number of episodes of hypernatremia | daily during ICU stay or up to day 90
  Number of episodes of hypernatremia (serum sodium > 145 mmol/L) during ICU stay (or up to day 90, whichever occurs first)
Glasgow coma scale at ICU and hospital discharge | at ICU discharge and hospital discharge
  Glasgow coma scale at ICU and hospital discharge
Number of patients with an episode of stroke | daily during ICU stay or up to day 90
  Number of patients with an episode of stroke (medical diagnosis as registered in the medical file) during ICU stay (or up to day 90, whichever occurs first)
Gastroduodenal bleeding | daily during ICU stay or up to day 90
  Gastroduodenal bleeding requiring transfusion or hemostatic treatment during ICU stay (or up to day 90, whichever occurs first)
Adult cognitive function score | at 1, 28, 90 day and 6 months
  Neurological cognitive dysfunction defined as by low score on the PROMIS (Adult cognitive function score).
  PROMIS (Patient-Reported Outcomes Measurement Information System): for assessment of fatigue, ability to partake in social activities, physical function, emotional distress, depression, anxiety and cognitive function.

CONTACTS AND LOCATIONS:
Overall Officials: Djillali ANNANE, MD, PhD, Principal Investigator — Department of medical and surgical Intensive Care Unit, - Raymond Poincaré Hospital - APHP
Locations (1):
- Department of medical and surgical Intensive Care Unit, Raymond Poincaré Hospital - APHP, Garches, Hauts-de-Seine, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Annane D, Pastores SM, Rochwerg B, Arlt W, Balk RA, Beishuizen A, Briegel J, Carcillo J, Christ-Crain M, Cooper MS, Marik PE, Umberto Meduri G, Olsen KM, Rodgers S, Russell JA, Van den Berghe G. Guidelines for the diagnosis and management of critical illness-related corticosteroid insufficiency (CIRCI) in critically ill patients (Part I): Society of Critical Care Medicine (SCCM) and European Society of Intensive Care Medicine (ESICM) 2017. Intensive Care Med. 2017 Dec;43(12):1751-1763. doi: 10.1007/s00134-017-4919-5. Epub 2017 Sep 21. PMID 28940011
- [Background] Lamontagne F, Rochwerg B, Lytvyn L, Guyatt GH, Moller MH, Annane D, Kho ME, Adhikari NKJ, Machado F, Vandvik PO, Dodek P, Leboeuf R, Briel M, Hashmi M, Camsooksai J, Shankar-Hari M, Baraki MK, Fugate K, Chua S, Marti C, Cohen D, Botton E, Agoritsas T, Siemieniuk RAC. Corticosteroid therapy for sepsis: a clinical practice guideline. BMJ. 2018 Aug 10;362:k3284. doi: 10.1136/bmj.k3284. No abstract available. PMID 30097460
- [Background] Rochwerg B, Oczkowski SJ, Siemieniuk RAC, Agoritsas T, Belley-Cote E, D'Aragon F, Duan E, English S, Gossack-Keenan K, Alghuroba M, Szczeklik W, Menon K, Alhazzani W, Sevransky J, Vandvik PO, Annane D, Guyatt G. Corticosteroids in Sepsis: An Updated Systematic Review and Meta-Analysis. Crit Care Med. 2018 Sep;46(9):1411-1420. doi: 10.1097/CCM.0000000000003262. PMID 29979221
- [Background] Nishida O, Ogura H, Egi M, Fujishima S, Hayashi Y, Iba T, Imaizumi H, Inoue S, Kakihana Y, Kotani J, Kushimoto S, Masuda Y, Matsuda N, Matsushima A, Nakada TA, Nakagawa S, Nunomiya S, Sadahiro T, Shime N, Yatabe T, Hara Y, Hayashida K, Kondo Y, Sumi Y, Yasuda H, Aoyama K, Azuhata T, Doi K, Doi M, Fujimura N, Fuke R, Fukuda T, Goto K, Hasegawa R, Hashimoto S, Hatakeyama J, Hayakawa M, Hifumi T, Higashibeppu N, Hirai K, Hirose T, Ide K, Kaizuka Y, Kan'o T, Kawasaki T, Kuroda H, Matsuda A, Matsumoto S, Nagae M, Onodera M, Ohnuma T, Oshima K, Saito N, Sakamoto S, Sakuraya M, Sasano M, Sato N, Sawamura A, Shimizu K, Shirai K, Takei T, Takeuchi M, Takimoto K, Taniguchi T, Tatsumi H, Tsuruta R, Yama N, Yamakawa K, Yamashita C, Yamashita K, Yoshida T, Tanaka H, Oda S. The Japanese Clinical Practice Guidelines for Management of Sepsis and Septic Shock 2016 (J-SSCG 2016). Acute Med Surg. 2018 Feb 5;5(1):3-89. doi: 10.1002/ams2.322. eCollection 2018 Jan. PMID 29445505
- [Background] Rhodes A, Evans LE, Alhazzani W, Levy MM, Antonelli M, Ferrer R, Kumar A, Sevransky JE, Sprung CL, Nunnally ME, Rochwerg B, Rubenfeld GD, Angus DC, Annane D, Beale RJ, Bellinghan GJ, Bernard GR, Chiche JD, Coopersmith C, De Backer DP, French CJ, Fujishima S, Gerlach H, Hidalgo JL, Hollenberg SM, Jones AE, Karnad DR, Kleinpell RM, Koh Y, Lisboa TC, Machado FR, Marini JJ, Marshall JC, Mazuski JE, McIntyre LA, McLean AS, Mehta S, Moreno RP, Myburgh J, Navalesi P, Nishida O, Osborn TM, Perner A, Plunkett CM, Ranieri M, Schorr CA, Seckel MA, Seymour CW, Shieh L, Shukri KA, Simpson SQ, Singer M, Thompson BT, Townsend SR, Van der Poll T, Vincent JL, Wiersinga WJ, Zimmerman JL, Dellinger RP. Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock: 2016. Intensive Care Med. 2017 Mar;43(3):304-377. doi: 10.1007/s00134-017-4683-6. Epub 2017 Jan 18. PMID 28101605
- [Background] Tavare A, O'Flynn N. Recognition, diagnosis, and early management of sepsis: NICE guideline. Br J Gen Pract. 2017 Apr;67(657):185-186. doi: 10.3399/bjgp17X690401. No abstract available. PMID 28360070
- [Background] van der Poll T, van de Veerdonk FL, Scicluna BP, Netea MG. The immunopathology of sepsis and potential therapeutic targets. Nat Rev Immunol. 2017 Jul;17(7):407-420. doi: 10.1038/nri.2017.36. Epub 2017 Apr 24. PMID 28436424
- [Background] Wong HR, Cvijanovich NZ, Anas N, Allen GL, Thomas NJ, Bigham MT, Weiss SL, Fitzgerald J, Checchia PA, Meyer K, Shanley TP, Quasney M, Hall M, Gedeit R, Freishtat RJ, Nowak J, Shekhar RS, Gertz S, Dawson E, Howard K, Harmon K, Beckman E, Frank E, Lindsell CJ. Developing a clinically feasible personalized medicine approach to pediatric septic shock. Am J Respir Crit Care Med. 2015 Feb 1;191(3):309-15. doi: 10.1164/rccm.201410-1864OC. PMID 25489881
- [Background] Antcliffe DB, Burnham KL, Al-Beidh F, Santhakumaran S, Brett SJ, Hinds CJ, Ashby D, Knight JC, Gordon AC. Transcriptomic Signatures in Sepsis and a Differential Response to Steroids. From the VANISH Randomized Trial. Am J Respir Crit Care Med. 2019 Apr 15;199(8):980-986. doi: 10.1164/rccm.201807-1419OC. PMID 30365341
- [Background] Annane D, Pastores SM, Arlt W, Balk RA, Beishuizen A, Briegel J, Carcillo J, Christ-Crain M, Cooper MS, Marik PE, Meduri GU, Olsen KM, Rochwerg B, Rodgers SC, Russell JA, Van den Berghe G. Critical illness-related corticosteroid insufficiency (CIRCI): a narrative review from a Multispecialty Task Force of the Society of Critical Care Medicine (SCCM) and the European Society of Intensive Care Medicine (ESICM). Intensive Care Med. 2017 Dec;43(12):1781-1792. doi: 10.1007/s00134-017-4914-x. Epub 2017 Sep 21. PMID 28940017
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] ARDS Definition Task Force; Ranieri VM, Rubenfeld GD, Thompson BT, Ferguson ND, Caldwell E, Fan E, Camporota L, Slutsky AS. Acute respiratory distress syndrome: the Berlin Definition. JAMA. 2012 Jun 20;307(23):2526-33. doi: 10.1001/jama.2012.5669. PMID 22797452
- [Derived] Fleuriet J, Heming N, Meziani F, Reignier J, Declerq PL, Mercier E, Muller G, Colin G, Monnet X, Robine A, Siami S, Uhel F, Quenot JP, Plantefeve G, Badie J, Schneider F, Cerf C, Troche G, Monchi M, Mira JP, Francois B, Chevret S, Annane D; RECORDS consortium; CRICS TRIGGERSEP network. Rapid rEcognition of COrticosteRoiD resistant or sensitive Sepsis (RECORDS): study protocol for a multicentre, placebo-controlled, biomarker-guided, adaptive Bayesian design basket trial. BMJ Open. 2023 Mar 10;13(3):e066496. doi: 10.1136/bmjopen-2022-066496. PMID 36898751